CLINICAL TRIAL: NCT06997224
Title: Comparison of the Effects of Triflow and Deep Breathing and Cough Exercises on Postoperative Respiratory Functions in Patients Undergoing Mitral Valve Replacement: A Randomized Controlled Trial
Brief Title: Effects of Triflow and Deep Breathing and Cough Exercises on Respiration in Patients Undergoing Mitral Valve Replacement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Cagla Toprak, Principal Investigator, Atlas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024-11
Record Dates: First submitted 2025-05-15; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Mitral Valve Failure; Surgery
Keywords: triflow; respiratory functions; cough exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- triflow group (Experimental): Before the operation, the experimental group will be taught the use of triflow and cough breathing exercises. On the first day after the operation, patients will be given triflow application 10 times every hour they are awake and cough and breathing exercises at other hours. Forms will be filled in before the application. After the application is completed at the end of the day, the forms will be filled in again. The application will continue until the patient is discharged.
  Interventions: Other: triflow application
- control group (No Intervention): After the surgery, patients will not be taught cough breathing exercises. Only the triflo application will be performed. The process will continue until discharge.

INTERVENTIONS:
Other: triflow application — After we have exhaled, we will try to hold the balls up as long as possible by pulling them inward with all our strength. After repeating this five times, we will turn them over.
  Arms: triflow group

SUMMARY:
The purpose of breathing exercises or the use of assistive devices is to provide deep breathing after surgery and to obtain a normal breathing pattern. The purpose of choosing the method to be applied is to obtain the best result. The results of the few studies conducted on this subject are contradictory and insufficient. In this context, the purpose of this study is to compare the effects of using only triflow and using triflow together with deep breathing and cough exercises on postoperative respiratory functions in patients who underwent simultaneous tricuspid valve surgery for mitral valve.

DETAILED DESCRIPTION:
Mitral valve disease is one of the most common causes of heart failure and death. Although heart valve diseases are not as common as heart failure, coronary artery disease or hypertension in developed countries, they are important because they are common and usually require intervention. In addition, rheumatic valve diseases are still an important public health problem in developing countries, and they mostly affect young patients. Since mitral valve diseases can progress without symptoms for a long time, when they are noticed, the damage to the valve may have reached a moderate or severe level. Therefore, it is necessary to carefully decide whether medical or surgical treatment is appropriate. The most common complications after mitral valve replacement are bleeding due to anticoagulant use, thromboembolism and deterioration in the valve structure, and some complications can be seen after surgery. The most common complications encountered are lung complications. The visibility of lung complications usually varies between 8-79%. The aim of this study is to compare the effects of using Triflow alone and using Triflow with deep breathing and cough exercises on postoperative respiratory functions in patients undergoing coronary artery bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study Literate and knowing the native language

Exclusion Criteria:

* Hemodynamically unstable patients, Patients who develop postoperative respiratory complications, Lip or palate anomalies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
The Visual Analog Scale (VAS) | perioperative 1 hour
  VAS is a one-dimensional scale used to measure subjective parameters. It consists of a 10-cm- long line drawn vertically or horizontally. At either end of this line are the two extreme descriptive words of the subjective category (0 = "no pain at all", 10 = worst/unbearable pain"). The patient is asked to indicate the point which matches his/her situation by placing a dot or drawing a line on this 10-cm-long line. It has been widely accepted in the world literature as a valid and reliable measurement tool in the evaluation of postoperative acute pain intensity.
The Visual Analog Scale (VAS) | postoperative evening
  VAS is a one-dimensional scale used to measure subjective parameters. It consists of a 10-cm- long line drawn vertically or horizontally. At either end of this line are the two extreme descriptive words of the subjective category (0 = "no pain at all", 10 = worst/unbearable pain"). The patient is asked to indicate the point which matches his/her situation by placing a dot or drawing a line on this 10-cm-long line. It has been widely accepted in the world literature as a valid and reliable measurement tool in the evaluation of postoperative acute pain intensity.
Postoperative Patient Follow-Up and Evaluation Form | postoperative evening
  It was created by researchers to evaluate cardiovascular and respiratory parameters, time to first mobilization, pain and complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akinci N, Eren E. Effects of combined Triflow, deep breathing and coughing exercises on postoperative pulmonary function after mitral valve replacement: a randomized controlled trial. BMC Surg. 2026 Feb 10. doi: 10.1186/s12893-026-03542-7. Online ahead of print. PMID 41668083